CLINICAL TRIAL: NCT04189549
Title: Preclinical Detection of Sepsis Early in Hospitalized Patients Following Surgery, Injury or Severe Illness (Pre-SEPSIS Trial)
Brief Title: Preclinical Detection of Sepsis Early in Hospitalized Patients Following Surgery, Injury or Severe Illness
Acronym: Pre-SEPSIS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Robert Ehrman (Other)
Responsible Party: Sponsor-Investigator, Robert Ehrman, Assistant Professor of Emergency Medicine, Wayne State University
Organization: Wayne State University (Other)
Other Study IDs: 2019R110
Record Dates: First submitted 2019-12-02; First posted 2019-12-06 (Actual); Last update posted 2019-12-06 (Actual); Status verified 2019-12

CONDITIONS: Sepsis
Keywords: Biomarker; Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Diagnostic Test: CNA Rapid Sepsis Dx — Novel biomarker based on circulating cell-free DNA (cfDNA) in the human blood stream

SUMMARY:
This clinical study is to evaluate a novel biomarker - CNA Rapid Sepsis Dx - to predict the development of sepsis in patients admitted to the hospital with non-sepsis conditions. Using circulating cell-free DNA (cfDNA) in the blood stream, it has been demonstrated to detect infection response days before clinical evidence of sepsis manifests. The hypothesis is that blood biomarkers drawn daily in the hospital will identify patients who develop sepsis within seven days of hospital presentation.

DETAILED DESCRIPTION:
This is a prospective observational trial evaluating CNA Rapid Sepsis Dx -novel biomarkers (CNA Diagnostics Inc.; Calgary, Canada) based on circulating cell-free DNA (cfDNA) in the blood stream to identify patients originally admitted with non-sepsis conditions who ultimately develop sepsis according to Sepsis-3 criteria within seven days of hospital presentation. This novel technology has been demonstrated to detect host-related response to infection days before clinical evidence of sepsis manifests.

The primary objective of this study is to assess the performance of the novel diagnostic assay, CNA Rapid Sepsis Dx, based on the biomarkers, drawn daily from the day of hospital presentation, to identify patients who ultimately develop sepsis according to Sepsis-3-definition within seven days of hospital presentation.

The secondary objective is to correlate the CNA Rapid Sepsis Dx with clinically relevant outcomes such as infections that otherwise do not meet Sepsis-3 criteria, intensive care unit (ICU) length of stay, hospital length of stay, fluid culture results, and hospital mortality.

ELIGIBILITY:
Inclusion Criteria:

1. Patient 18 years of age or older at the time of enrollment
2. Presence of any of the following high-risk features:

   * Victims of trauma with either an Injury Severity Score of ≥ 15 or a Glasgow Coma Score of ≤ 8[2] OR
   * Any patient undergoing high-risk surgical procedures including any emergency surgery and high risk elective surgery procedures involving the thorax, esophagus, stomach, small bowel, large bowel [3, 4] OR
   * Any patient being admitted to any ICU setting for any reason with no current evidence or suspicion of active infection (by primary team).[5, 6]
3. Able to collect sample within 24 hours of presentation to the hospital.

Exclusion Criteria:

1. Prisoners or in police custody
2. Pregnancy
3. Pre-existing infection for which patient is being treated with antibiotics as an outpatient.
4. Plan for ongoing antibiotic therapy by treating team (up to three doses antibiotics for peri-procedure prophylaxis is allowable).
5. Moribund, unlikely to survive the duration of active enrollment
6. Comfort care measures in place or ordered at time of screening OR indication from treating team that active medical care will not be pursued due to patient's condition or patient's/family's wishes.
7. Palliative care or hospice consult at time of screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the hospital and admitted for non-sepsis conditions who are at increased risk for developing sepsis per Sepsis-3 criteria within the hospital.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2019-12-09 (Estimated); Primary Completion 2020-11-01 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
Clinical development of sepsis | Seven Days from hospital presentation
  Sepsis determined according to Sepsis-3 definition

SECONDARY OUTCOMES:
SIRS sepsis | Seven Days from hospital presentation
  Infection with systemic inflammatory response syndrome (SIRS) criteria
Hospital Length of Stay | Up to 12 months
  Duration of hospital stay in survivors and non-survivors from date/time of hospital presentation to order for discharge.
Intensive Care Unit Length of Stay | Up to 6 months
  Duration of ICU stay in survivors and non-survivors from date/time of ICU admission to date/time order for transfer / discharge from ICU.
Development of non-Sepsis 3 Infections | Seven Days from hospital presentation
  An infection is suspected (by any degree of confidence) but the subject does not meet criteria for either Sepsis-3 or SIRS sepsis.
Body Fluid Culture Results | Seven Days from hospital presentation
  All fluid culture results (blood, CSF, urine, synovial, ascitic, abscess, etc) collected during the study period will be recorded

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - University of Alabama Birmingham, Birmingham, Alabama
  - Detroit Receiving Hospital, Detroit, Michigan
  - Harper University Hospital, Detroit, Michigan
  - Sinai-Grace Hospital, Detroit, Michigan
  - Northwell Health, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided